CLINICAL TRIAL: NCT01885390
Title: ROX CONTROL HTN Registry: To Evaluate the ROX Coupler in Patients With Resistant or Uncontrolled Hypertension
Brief Title: Registry to Evaluate the ROX COUPLER in Patients With Resistant or Uncontrolled Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ROX Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RH-03
Record Dates: First submitted 2013-06-20; First posted 2013-06-25 (Estimated); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: Hypertension; Blood Pressure, High; Blood Pressure, Resistant; Blood Pressure, Uncontrolled
Keywords: Hypertension; High blood pressure; Resistant blood pressure; Uncontrolled blood pressure
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental: Group A (Experimental): ROX Coupler + continuing standard antihypertensive medications
  Interventions: Device: ROX COUPLER

INTERVENTIONS:
Device: ROX COUPLER — The COUPLER will be used to create an anastomosis in the iliac region (between the iliac artery and vein).

SUMMARY:
The purpose of this registry is to evaluate the safety and performance of the ROX COUPLER in patients with treatment-resistant or uncontrolled hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of resistant or uncontrolled hypertension must be made on the basis of current findings, medical history, and physical examination.

Exclusion Criteria:

* Any serious medical condition that may adversely affect the patient's safety, limit the subject's ability to participate in the registry, comply with follow-up requirements, or impact the scientific integrity of the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2019-05-05 (Actual); Study Completion 2019-05-05 (Actual)

PRIMARY OUTCOMES:
Change in ambulatory daytime mean systolic blood pressure | Baseline, 6 months
  Change in mean ambulatory daytime systolic blood pressure at six months as compared to Baseline.

SECONDARY OUTCOMES:
Change in ambulatory daytime mean diastolic blood pressure | Baseline, 6 months
  Change in mean ambulatory daytime diastolic blood pressure at six months as compared to Baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Mel Lobo, MD, Principal Investigator — Queen Mary University of London
Locations (4):
- ZNA Cardio Middelheim, Antwerp, Belgium
- St. Antonius Ziekenhuis, Nieuwegein, Netherlands
- United Kingdom (2):
  - East Sussex Healthcare NHS Trust, Eastbourne
  - Queen Mary University of London, London